CLINICAL TRIAL: NCT07329621
Title: A Phase 1, Open-label, Positron Emission Tomography (PET) Trial to Measure Serotonin 5-HT2A Receptor Occupancy Following Single Oral Doses of MSP-2020 in Healthy Male Adults
Brief Title: A Brain Imaging Study to Assess the Binding of MSP-2020 to Serotonin 5-HT2A Receptors in Healthy Male Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 358-201-00002
Record Dates: First submitted 2025-12-19; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Incomplete Response - Major Depressive Disorder (IR-MDD)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MSP-2020 Oral Administration (Experimental): Participants will receive a single dose of MSP-2020 on Day 1.
  Interventions: Drug: MSP-2020

INTERVENTIONS:
Drug: MSP-2020 — capsule

SUMMARY:
This study is to see how well MSP-2020 attaches to specific targets in the brain called serotonin type 2A receptors (5-HT2AR). This study will also look at how much of the study drug (and its active metabolite) is in the blood and how long the study drug stays in the blood, as well as the safety of MSP 2020.

ELIGIBILITY:
Inclusion Criteria

1. Able to stay in the CRU for up to 4 days.
2. Body mass index (BMI) between 18.0 to 32.0 kg/m2 (inclusive).
3. In good health as determined by: a. Medical history; b. Physical and neurological examination; c. Concomitant medications; d. ECG; e. Screening echocardiogram; f. Serum chemistry, urinalysis, haematology, coagulation, and serology (HIV screen, HBsAg, and anti-HCV) tests.

Exclusion Criteria

1. In first-degree relatives, a history of any schizophrenia-spectrum disorder, psychotic disorder, or bipolar and related disorders.
2. History of allergy to tracer [11C]CIMBI-36.
3. MRI incompatibility due to implants including but not limited to pacemaker, artificial joints, or non-removable body piercings, and/or other contraindications for MRI such as claustrophobia, metal objects/fragments, or fragments in the head or body that would present a risk during the MRI scanning procedure, or have worked with ferrous metals (eg, welding), or have motor problems that prevent the participant from lying still for the MRI.
4. Pathological MRI findings that would preclude from trial participation.
5. History of prior radiation exposure for research purposes such that participation in this trial would result in an ionising radiation exposure of > 10 mSv within a year (12 months) of the first PET scan that would cause the participant to exceed the yearly dose limit.
6. Have a negative modified Allen test at screening.
7. Contraindications to radial arterial cannula (including but not limited to cellulitis or other infections over the radial artery, absence of palpable radial artery pulse, or a clinically significant abnormal coagulation profile).
8. Clinically significant abnormality in past medical history, or at the screening physical examination, that in the investigator's or sponsor's opinion may place the participant at risk or interfere with outcome variables including absorption, distribution, metabolism, and excretion of drug. This includes, but is not limited to, history of or concurrent cardiac, hepatic, renal, neurologic, endocrine, gastrointestinal, respiratory, haematologic, dermatologic, and immunologic disease.
9. History of alcohol and/or substance use disorder within the last 24 months according to the Diagnostic Statistical Manual of Mental Disorders and in past medical history or in the investigator's opinion, or intake of > 21 units of alcohol weekly, and the inability to refrain from alcohol use from 48 hours before screening and within 72 hours prior to dosing until discharge from the CRU on Day 2. One unit is equivalent to 1 (25 mL) measure of 40% spirits. For reference, one 330 mL bottle of 5% beer contains 1.7 units and a standard (175 mL) glass of 12% wine contains 2.1 units.

Note: Other protocol-specified Inclusion/Exclusion criteria may apply.

Ages: 23 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-10-12 (Estimated); Study Completion 2026-10-25 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Specific Binding of [11C]CIMBI-36 from Baseline and EC50 Using Cortical Regions [11C]CIMBI-36 BPND | Up to Day 2
PK Plasma Concentration of MSP-2020 and its Metabolite | Up to Day 2
Maximum (peak) Plasma Concentration of MSP-2020 and its Metabolite | Up to Day 2
Time to Maximum (peak) Plasma Concentration of MSP-2020 and its Metabolite | Up to Day 2
Half-life (t1/2) of MSP-2020 and its metabolite | Up to Day 2
Area under the concentration-time curve (AUCt) of MSP-2020 and its metabolite | Up to Day 2

SECONDARY OUTCOMES:
Change from Baseline in Subjective Drug Intensity Scale Score | Up to Day 2
Change from Baseline in 5-Dimensional Altered States of Consciousness (5D-ASC) Score | Up to Day 2
Change from Baseline in 30-item Mystical Experience Questionnaire (MEQ-30) Score | Up to Day 2
Change from Baseline in Ego-Dissolution Inventory (EDI) Score | Up to Day 2
Concentration of the metabolite at which 50% of the 5-HT2A receptors are occupied, as measured by PET imaging | Up to Day 2
Number of Participants With Adverse Events (AEs) | Up to Day 15
Number of Participants With Potentially Clinically Significant Changes in Vital Signs | Up to Day 2
Number of Participants With Potentially Clinically Significant Changes in Electrocardiogram (ECG) | Up to Day 2
Number of Participants With Potentially Clinically Significant Changes in Laboratory Tests | Up to Day 15
Number of Participants With Potentially Clinically Significant Changes in Physical and Neurological Examinations | Up to Day 15
Number of Participants With Suicidality on Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- HMR Hammersmith Medicines Research Ltd., London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymized individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.